CLINICAL TRIAL: NCT06440109
Title: The Effect of Therapeutic Touch and Emotional Freedom Technique on Postpartum Mood and Fatigue in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A-TURAN-001
Record Dates: First submitted 2024-05-08; First posted 2024-06-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-03

CONDITIONS: Fatigue; Emotion Regulation
Keywords: emotional freedom technic; therapeutic touch; fatigue; mood state level
MeSH Terms: conditions — Fatigue; Emotional Regulation | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EFT intervention (Experimental): The application will be carried out in line with EFT application protocols. In this regard, women's home visits will be completed with 6 meetings, once every week. Each EFT session will last 15 minutes
  Interventions: Other: Emotional freedom technique (EFT)
- TD intervention (Experimental): The application will be carried out in line with TD application protocols. In this regard, women's home visits will be completed with 6 meetings, once every week. Each TD session will last 15 minutes
  Interventions: Other: Therapeutic touch (TD)
- Control grup (No Intervention): No intervention will be made. Women in the intervention groups will be followed for 6 weeks and receive standard care. The final test will be administered at the end of the sixth week

INTERVENTIONS:
Other: Emotional freedom technique (EFT) — İntervention groups will be followed for six months and one of the six EFT therapies will be applied, one session every week.
  Arms: EFT intervention
Other: Therapeutic touch (TD) — İntervention groups will be followed for six weeks and one of the six TD therapies will be applied, one session every week.
  Arms: TD intervention

SUMMARY:
Therapeutic touch (TD) is a non-pharmacological/integrated treatment method used to balance the body by regulating the imbalanced energy field in the individual or resolving blockages in energy flow. Emotional freedom technique (EFT) is a psychophysiological intervention that combines elements of somatic stimulation using acupuncture points. This research will be conducted as a randomized controlled experimental study to determine the effect of TD and EFT intervention on postpartum mood and fatigue in postpartum women. This study is planned to be conducted between April 2024 and June 2025 with postpartum women who meet the inclusion criteria and who apply to the Obstetrics and Gynecology Clinic of Necmettin Erbakan University Faculty of Medicine Hospital. This research; It was planned to be carried out with three groups: TD intervention, EFT intervention and control group. The population of the research consists of women who gave birth vaginally and those who gave birth vaginally in the relevant hospital.

ELIGIBILITY:
Inclusion Criteria:

* Having a vaginal birth at term
* Being primiparous
* Postpartum 3rd-5th. to be in the days
* Being able to speak and understand Turkish
* Being 18 years or older
* Having a single and viable fetus
* Volunteering to participate in research
* Not having experienced TD or EFT treatment before

Exclusion Criteria:

* A psychiatric diagnosis has been made,
* Having a chronic systemic disease,
* The newborn's need for treatment
* Having postpartum complications in the mother or baby
* Those who have sensitivity or problems with touch,
* Wounds, infections, etc. in places that need to be touched. existence of situations,
* Women who have any disability that would prevent communication (deafness, hearing impairment, etc., use of languages other than Turkish) will be excluded from the research.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Postpartum 1rd-5th. EFT intervention will be applied to women who are between | six weeks
  SUE scale and vital signs will be taken from the participants before and after each session.
Postpartum 3rd-5th. TD intervention will be applied to women who are between | six weeks
  SUE scale and vital signs will be taken from the participants before and after each session.
3rd-5th postpartum Pre- and post-test will be given to women between | six weeks
  The researcher will not perform any intervention on women in this group. After the pre-tests are completed, women in this group will be called by phone during the interview weeks for the intervention group, their postpartum needs will be questioned and support will be provided when necessary. The implementation of the final tests will be completed in the sixth week.

CONTACTS AND LOCATIONS:
Overall Officials: Aslıhan Turan, PhD (c), Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No